CLINICAL TRIAL: NCT05636254
Title: Diagnostic Accuracy of Imaging Findings in Tubercular Meningitis/Spinal Tubercular Arachnoiditis and Correlation With Outcomes in Patients With Tubercular Meningitis, Spinal Tubercular Arachnoiditis
Brief Title: Diagnostic Accuracy of Imaging Findings in TBM/Spinal Tubercular Arachnoiditis and Correlation With Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Assistant Professor of Neurology, All India Institute of Medical Sciences
Other Study IDs: IECPG-36/27.01.2022
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Tuberculous Meningitis; Tuberculous Arachnoiditis
Keywords: TBM
MeSH Terms: conditions — Tuberculosis, Meningeal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Meningitis: * Chronic meningitis : Case definition
    * Headache with or without fever, nuchal stiffness and systemic symptoms AND
    * CSF suggestive of meningitis Pleocytosis (>20 cells per μL) with lymphocyte predominance (>50%) OR Protein concentration greater than age-specific normal value; especially >1•0 g/L OR Glucose concentration less than 60% of concentration in blood OR MRI suggestive of meningeal enhancement on contrast enhanced T1 sequences AND
    * Deemed by the treating physician that the syndrome is consistent with chronic meningitis
  * Patients who are positive for antibodies to HIV and pregnant females will also be included.
  Interventions: Diagnostic Test: MRI Brain and spine; Diagnostic Test: Reference standard diagnostic criteria

INTERVENTIONS:
Diagnostic Test: MRI Brain and spine — * MRI Brain
  * Ax T2 TSE
  * 3D Sag T1
  * Ax DWI
  * 3D Sag Flair
  * Ax SWI
  * Post-gad 3D Sag T1
  * 3D TOF Circle-of-Willis
  * MRI Spine
  * Sag T2 whole spine (2 stations)
  * Post-gad Sag T1 whole spine (2 stations)
Diagnostic Test: Reference standard diagnostic criteria — Diagnostic criteria-TBM
  * Microbiologic evidence of TB in CSF
  * Microbiologic evidence of TB from pulmonary or extrapulmonary sites
  * Reasonable clinical certainty OR allied investigations such as CXR/CECT chest/abdomen/PET CT as per clinical indication suggestive of tuberculosis
  * Other relevant investigations like CSF analysis not suggestive of alternative diagnosis such as neurocysticercosis/cryptococcal/other fungal infections/other causes of chronic meningitis such as brucella/ nocardia/ syphilis/recurrent viral meningitis/ carcinomatous/ lymphomatous meningitis or non infective causes such as sarcoidoisis/sub-arachnoid hemorrhage etc.
  * Reasonable clinical certainty OR allied investigations such as CXR/CECT chest/abdomen/PET CT as per clinical indication ruling out competing diagnoses
  * Patients who develop features or test results suggestive of alternative diagnosis with will be considered to be not due to tubercular meningitis
  Other Names: Clinical composite criteria

SUMMARY:
The goal of this Diagnostic accuracy study is

* To study sensitivity and specificity of sulcal tuberculomas in the diagnosis of tubercular meningitis and
* To study the correlation of imaging findings in tubercular meningitis and spinal tubercular arachnoiditis with clinical outcomes after completion of therapy
* Secondary objectives
* To study the proportion of patients having clinical or imaging features of spinal tubercular arachnoiditis
* To study the factors determining outcomes in patients with spinal tubercular arachnoiditis
* To study the treatment trends in patients with spinal tubercular arachnoiditis

The investigators will include [study Population] Patients with chronic meningitis as per criteria listed below

* Chronic meningitis : Case definition
* Headache with or without fever, nuchal stiffness and systemic symptoms AND
* CSF suggestive of meningitis Pleocytosis (>20 cells per μL) with lymphocyte predominance (>50%) OR Protein concentration greater than age-specific normal value; especially >1•0 g/L OR Glucose concentration less than 60% of concentration in blood OR MRI suggestive of meningeal enhancement on contrast enhanced T1 sequences AND
* Deemed by the treating physician that the syndrome is consistent with chronic meningitis
* Patients who are positive for antibodies to HIV and pregnant females will also be included.
* Willing to undergo periodic assessment clinically and with MRI as per clinical condition demands.

The sensitivity and specificity of the finding of sulcal tuberculomas will be compared to the reference standard diagnostic criteria for the diagnosis of TB meningitis.

DETAILED DESCRIPTION:
Methodology of the study Study design:Ambispective cohort study; Observational study; Diagnostic accuracy study

Sample size: All consecutive patients in the database will be included in the retrospective study and all new patients registered in the neurology OPD and admitted in the Neurology or General Medicine or Geriatric medicine or Medical oncology wards will be included in the prospective arm

Expecting a sensitivity of 70% of sulcal tuberculomas in tubercular meningitis with a range of 60 to 80, the investigators expect (4*70*30) /10*10=84 patients Expecting sulcal tuberculomas to have a specificity of 80%, with a range of 70 to 90%, the investigators expect (4*80*20)/10*10=64 patients Expecting a 70% prevalence of tubercular meningitis amongst patients with chronic meningitis, sample size of atleast 120 patients (70% of 120=84).

Subjects:

* Study Population: Patients with chronic meningitis as per criteria described
* Inclusion criteria

  * Patients attending Neurology OPD or are admitted in General Medicine or Geriatric medicine or Medical oncology wards with chronic meningitis diagnosed on the basis of composite clinical criteria, imaging criteria as well as natural history of the illness
  * Atleast 14 years of age of all sexes
  * Chronic meningitis : Case definition above
  * Willing to undergo periodic assessment clinically and with MRI as per clinical condition demands.
* Diagnostic criteria for Tuberculous meningitis ▪ Described in the diagnostic test section ahead
* Diagnostic criteria for clinical spinal tubercular arachnoiditis

  ▪ Developed paraparesis/quadriparesis/sphincter dysfunction due to spinal radiculomyelitis OR areflexia OR hyperreflexia with no obvious brain parenchymal lesions (suggestive of spinal meningitis-myelitis) or vision loss due to optico-chiasmatic arachnoiditis with imaging evidence of arachnoiditis
* Sample Size: All consecutive patients presenting with chronic meningitis as described above will be included

Exclusion criteria for prospective arm

● Not willing to provide consent

Conduct of the study

* Study protocol

  * Consent: Participants or their legally authorized representatives will be explained about the study and informed written consent will be taken in the language they understand for the prospective study
  * Participants will undergo magnetic resonance imaging of the brain and spine with contrast using the standardized protocol for chronic meningitis used at AIIMS as the standard of care in the workup of chronic meningitis.
  * The final diagnosis of Tubercular meningitis will be made based on the criteria described above and the sensitivity and specificity of sulcal tuberculomas in the diagnosis of TBM will be determined
  * Other imaging findings of spinal tubercular arachnoiditis will be collected on a structured proforma by the radiologist who will be blinded to the clinical information on the presence or absence of clinical features.
  * Participants will follow treatment for tuberculosis as per the treating physician's discretion in terms of anti-tubercular therapy, anti-seizure medication therapy, duration and dose of corticosteroids and steroid sparing agents.
  * Data collection and analysis will be done as per protocol Follow up and outcomes assessed > Participants of the prospective arm will be carefully assessed with detailed history, clinical examination, necessary laboratory investigations and imaging > Detailed history and clinical and neurologic examination, lab parameters and imaging data will be documented into a database as per protocol > Participants will follow treatment for his/her primary condition as per the treating physician's discretion > Outcomes will be assessed at 3 months, 6 months and at end of therapy > The outcome parameters of interest will be modified Rankin scale, visual acuity at 3 months and end of therapy.

Diagnostic accuracy of imaging parameters in the diagnosis of tubercular meningitis will be assessed by sensitivity and specificity.

The investigators aim to do a descriptive study of the clinical, laboratory and imaging parameters of patients tubercular meningitis and spinal tubercular arachnoiditis and compare with patients with other forms of chronic meningitis.

The treatment strategy, usage of anti-tubercular therapy, usage of corticosteroids, steroid sparing therapy, and surgical interventions offered will be studied.

Outcomes will be assessed and compared those who have sulcal tuberculumas and those who don't. The patients with and without spinal arachnoiditis on imaging also will be compared, and their outcomes assessed. Factors affecting outcomes will be studied and exploratory analysis will be done. Statistical analysis will be performed on the available information. Qualitative data will be presented as the number and the percentage of patients in each treatment group. Quantitative data will be presented as mean and standard deviation, range, median and inter-quartile range by treatment group. The absence of imbalance between groups will be checked on baseline variables. Comparisons of qualitative variables between groups will be performed by a Fisher exact test; comparison of quantitative data will be performed by a t test or a comparison of median when they will not follow a Normal distribution. All statistical tests will be performed with the use of a two-sided type I error rate of 5%.

ELIGIBILITY:
* Patients attending Neurology OPD or are admitted in General Medicine or Geriatric medicine or Medical oncologywards with chronic meningitis diagnosed on the basis of composite clinical criteria, imaging criteria as well as natural history of the illness
* Atleast 14 years of age of all sexes Willing to undergo periodic assessment clinically and with MRI as per clinical condition demands.

Exclusion Criteria:

Not willing to provide consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ▪ Chronic meningitis : Case definition
  * Headache with or without fever, nuchal stiffness and systemic symptoms AND
  * CSF suggestive of meningitis Pleocytosis (>20 cells per μL) with lymphocyte predominance (>50%) OR Protein concentration less greater than age-specific normal value; especially >1•0 g/L OR Glucose concentration than 60% of concentration in blood OR MRI suggestive of meningeal enhancement on contrast enhanced T1 sequences AND
  * Deemed by the treating physician that the syndrome is consistent with chronic meningitis
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of sulcal tuberculomas in the diagnosis of tubercular meningitis | Day 1 of diagnosis or imaging acquisition
  Sensitivity and specificity of sulcal tuberculomas compared with reference standard clinical composite criteria
Correlation of imaging findings with clinical outcomes | 6 months to 18 months, average 9 months after starting treatment
  Correlation of imaging findings in tubercular meningitis and spinal tubercular arachnoiditis with clinical outcomes after completion of therapy The outcome parameters of interest will be modified Rankin scale, visual acuity at 3 months and end of therapy.

SECONDARY OUTCOMES:
Clinical or imaging features of spinal tubercular arachnoiditis | Day 1 of diagnosis or imaging acquisition
  Proportion of patients having clinical or imaging features of spinal tubercular arachnoiditis
Factors determining outcomes in patients with spinal tubercular arachnoiditis | 6 months to 18 months, average 9 months after starting treatment
  Factors determining outcomes in patients with spinal tubercular arachnoiditis
Treatment trends in patients with spinal tubercular arachnoiditis | 6 months to 18 months, average 9 months after starting treatment
  Treatment trends in patients with spinal tubercular arachnoiditis

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
To be routed through proper channel through the ethics committee
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 3 months of request till five years after publication of results